CLINICAL TRIAL: NCT06000423
Title: Tranexamic Acid to Reduce Contraceptive-related Bleeding Side Effects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Alison Edelman, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OHSU IRB 25761
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Bleeding; Contraceptive Device; Complications
Keywords: Tranexamic Acid; Contraceptive Implant
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Participants assigned to either the TXA treatment group or the placebo group.
Who Masked: Participant, Investigator
Masking Description: double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): After three consecutive days of bleeding, five days of 1300mg TXA three times per day (TID).
  Interventions: Drug: Tranexamic acid
- Placebo (Placebo Comparator): After three consecutive days of bleeding, five days of placebo three times per day.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — 1300mg TXA taken three times per day for five days
  Other Names: TXA
  Arms: Treatment
Other: Placebo — Placebo pills taken three times daily for five days.
  Arms: Placebo

SUMMARY:
This randomized double blinded trial seeks to determine whether tranexamic acid (TXA) is an efficacious treatment for contraceptive induced menstrual changes (CIMC) including irregular, bothersome bleeding caused by the etonogestrel subdermal contraceptive implant (ENG implant). Participants will be randomized into the TXA treatment arm or a placebo. They will begin taking the medication after three consecutive days of bleeding. Participants will track their bleeding using an automated text message service

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* In good general health
* Have etonogestrel (ENG) subdermal contraceptive implant (must be palpable to prove that an ENG implant is in place at time of screening and enrollment)
* Experience frequent or prolonged bleeding while using ENG implant (>7 days of continuous bleeding/spotting in the last 30 days, or 2 or more episodes of bleeding/spotting in the last 30 days)
* Implant use for at least 30 days prior to screening visit
* Willing to continue using the implant for at least 30 days from study enrollment
* Access to a reliable cell phone and must be willing to receive and respond to a daily text or email message to assess bleeding and use of study drug
* Negative gonorrhea/chlamydia screening performed at screening visit

Exclusion Criteria:

* Centers for Disease Control Medical Eligibility for Contraceptive use category 3 or 4 for contraceptive usage
* Currently pregnant
* Less than 6 months postpartum, less than 6 weeks abortion, not breast/chest feeding (cessation of lactation at least 6 weeks prior to enrollment)
* Undiagnosed abnormal uterine bleeding pre-dating placement of contraceptive implant
* Bleeding dyscrasia
* Anticoagulation use
* Active cervicitis
* Allergy to Tranexamic Acid
* Known renal insufficiency
* History of venous thromboembolism
* Current or past breast or uterine malignancy
* Concurrent use of P450 pathway inducing drug
* Implant is due to be switched out in 2 months or less from enrollment
* Routine or chronic use of non-steroidal anti-inflammatory drugs (NSAIDs once daily or >= 14 days per month)
* Currently using oral contraceptives in addition to implant (to be eligible, needs to have 4-6 week washout period)
* Prior pregnancy occurred while Nexplanon/Implanon was in place
* Chronic use of Cannabidiol, THC, or marijuana (>3 times per week) (patients could have used Cannabidiol, THC, or marijuana chronically in the past, but must have a washout time period of no use for at least one month prior to the study)
* Chronic use of cigarettes (>1 cigarette per week) (patients could have used cigarettes chronically in the past, but must have a washout time period of no use for at least six months prior to the study)

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Amenorrhea days | 30 days
  The difference in mean days without bleeding across 30-day reference period between the treatment and placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Edelman, MD, MPH, Principal Investigator — Oregon Health and Science University; Leo Han, MD, MCR, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No